CLINICAL TRIAL: NCT01138683
Title: Cardiorenal Interactions During Treatment of Acute Decompensated Heart Failure: Diuretics Versus Ultrafiltration
Acronym: CRUF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/539; 2009-017589-22 (EudraCT Number)
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acute decompensated heart failure; ultrafiltration; diuretics; AKI
MeSH Terms: interventions — Ultrafiltration; Diuretics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultrafiltration group (Active Comparator)
  Interventions: Procedure: ultrafiltration
- diuretics group (Active Comparator)
  Interventions: Drug: diuretics

INTERVENTIONS:
Procedure: ultrafiltration — Ultrafiltration through double lumen catheter, via central vein (Vena jugularis interna or Vena femoralis, 11 French, 15 cm for right jugular or 20 cm for femoralis and jugularis left-position). Based on severity of fluid overload the cardiologist determines the ultrafiltration rate. 'Multifiltrate Fresenius' (extracorporeal blood volume 72ml) in SCUF (slow continuous ultrafiltration) modus with pediatric lines (54 ml extracorporeal volume in the AV-set) and a pediatric filter (Ultraflux® AV paed, blood volume 18ml). Heparin to maintain an APTT between 65 en 85 seconds during ultrafiltration.
  Arms: ultrafiltration group
Drug: diuretics — Bumetanide continuous infusion to reach a prescribed negative fluid balance: dose adjustment according to the diuretic response.
  Arms: diuretics group

SUMMARY:
The CRUF trial is a prospective randomized monocentric trial comparing different impact of diuretics versus ultrafiltration on renal congestion, plasma refill rate, echocardiographic filling pressures, neurohormonal activation and biomarkers of Acute Kidney Injury (AKI).

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Severe systolic heart failure with ejection fraction <40%
* And Hospitalisation for decompensated heart failure
* And New York Heart Association (NYHA) III or IV
* And 1 of the following:

  * Jugular vein distension>6cm
  * Tissue Doppler mitral annulus lateral>12 or medial>15
  * Chest X-ray: pulmonary edema or pleural effusion

Exclusion Criteria:

* Need for inotropic or vasopressive agents
* Use of intravenous (IV) contrast media
* Acute coronary syndrome
* Need of dialysis
* Severe co-morbidity
* Contra-indications for anticoagulation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI and determining factors in patients with acute decompensated heart failure with treated with ultrafiltration versus diuretics | at 6 months

SECONDARY OUTCOMES:
determination of the value of Neutrophil gelatinase-associated lipocalin (NGAL) to predict AKI in acute decompensated heart failure (vs creatinine, Cystatin C,measured urinary creatinine clearance) in patients treated with diuretics vs ultrafiltration. | at 48h after treatment start
Combined endpoint of mortality/rehospitalisation-urgent outpatient visit due to heart failure | at 6 months
Kidney function measured by creatinine | after 28 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Gevaert, MD, Principal Investigator — University Hospital Ghent, Belgium
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of University Hospital Ghent — http://www.uzgent.be